CLINICAL TRIAL: NCT02982538
Title: Implementation of Prolonged Exposure in the Army: Is Consultation Necessary for Effective Dissemination?
Brief Title: Implementation of Prolonged Exposure in the Military
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Texas (Other)
Responsible Party: Principal Investigator, Edna Foa, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: W81XWH-12-2-0116
Record Dates: First submitted 2016-01-25; First posted 2016-12-05 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: PTSD
Keywords: posttraumatic stress symptoms; implementation; dissemination; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard PE Training Condition (Other): Providers in this condition will complete a 4-day training workshop in PE.
  Interventions: Behavioral: Standard Training in Prolonged Exposure Therapy for PTSD
- Extended PE Training Condition (Other): Providers in this condition will complete a 4-day training workshop in PE and will receive expert PE case consultation on two PE training cases via weekly phone consultation.
  Interventions: Behavioral: Extended Training in Prolonged Exposure Therapy for PTSD

INTERVENTIONS:
Behavioral: Extended Training in Prolonged Exposure Therapy for PTSD — Extended training in Prolonged Exposure consists of a 4-day PE workshop, followed by expert PE consultation on 2 training cases. PE consultation consists of weekly telephone calls with expert PE therapists at the University of Pennsylvania, who will review video-recordings of providers PE sessions and provide feedback. Consultation is considered complete if the consultant has reviewed a minimum of 12 video-recorded sessions across 2 training cases, and has provided feedback on all of the crucial elements of PE (e.g., rationale, imaginal exposure, in vivo exposure, processing).
  Arms: Extended PE Training Condition
Behavioral: Standard Training in Prolonged Exposure Therapy for PTSD — Standard training in PE consists of a 4-day professional workshop on Prolonged Exposure Therapy. This is similar to the standard training approach that has been used to train providers in delivery of PE in the Army.
  Arms: Standard PE Training Condition

SUMMARY:
This randomized study examines how prolonged exposure (PE) therapy, an evidence-based treatment for posttraumatic stress disorder (PTSD), can be successfully disseminated and implemented in the Army. The study compares two PE training models: Standard PE training, comprised of a 4-day workshop only, and Extended PE training, comprised of a 4-day workshop plus expert case consultation. In addition, patients with posttraumatic stress symptoms receiving psychotherapy from participating providers will be invited to participate. After completing PE training, use of PE components with patients reporting PTS symptoms and clinical outcomes of these participating patients will be monitored for up to 18 months.

DETAILED DESCRIPTION:
This study will examine how evidence-based therapies (EBTs) such as Prolonged Exposure (PE) for posttraumatic stress disorder (PTSD) can be successfully disseminated and implemented in the Army by comparing two PE training models: Standard PE training (workshop only) and Extended PE training (workshop plus consultation). Up to 180 mental health providers at three medium-to large Army installations will be randomly assigned to either Standard PE training or Extended PE training. All providers will complete a 4-day PE workshop, along with the distribution of training materials and treatment manuals, conducted at the military site by the Overall Study PI, Dr. Edna Foa, and her team. Following the 4-day workshop, participants randomized to the Extended PE training will receive weekly phone consultation with a PE expert on two PE therapy cases. Participants randomized to the Standard PE training group will not receive any additional consultation following the workshop. Providers will not be required to use PE therapy with their patients with PTS symptoms; using PE will be optional. A major outcome of this study is the proportion of the providers PTSD patients that are offered PE or PE components. The mental health outcomes of providers' PTS patients will also be monitored as a second major outcome. Patients seeking treatment from participating providers will be recruited, consented, and assessed by independent evaluators at two time points to prospectively assess their response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* FOR PROVIDERS: 1) Male and female behavioral health providers whose job duties include providing psychotherapy to adult patients, age ≥ 18,seeking treatment with symptoms of PTS. Behavioral health providers can include psychologists, social workers, psychiatric clinical nurse specialists, psychiatrists, and similarly trained professional providers.2) Twenty percent (or more) of expected caseload comprised of patients with PTS symptoms according to provider self-report.
* FOR PATIENTS: 1) Male and female patients age ≥ 18. 2) Receiving treatment from one of the behavioral health providers participating in this study. 3) Significant PTS symptoms as determined by a score of 25 or higher on The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).

Exclusion Criteria:

* FOR PROVIDERS: 1) Definite plans to terminate their position or relocate from the Army base at some point during the first year following training. 2) Extensive previous training in Prolonged Exposure (PE), defined as participation in a 4-day PE training workshop at any point prior to the start of the study, and self-reported use of PE (including both imaginal and in vivo exposure techniques) to treat 4 or more patients with PTS symptoms in the past year.
* FOR PATIENTS: 1) Current bipolar disorder I or psychotic disorder (as determined by the MINI). 2) Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires). 3) Current suicidal ideation severe enough to warrant immediate attention (as determined by the MINI and the Beck Scale for Suicidal Ideation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Provider Use of PE Components | Through study completion, an average of 2 years
  Provider use of PE components will be assessed using a brief checklist of treatment procedures completed by providers directly following therapy sessions with participating patients.

SECONDARY OUTCOMES:
Provider Attitudes | Through study completion, an average of 2 years
  Provider change in self-efficacy and attitudes toward PE will be assessed via a self-report measure administered before and after the PE workshop, and at 3 month intervals until 18 months following the conclusion of training.
Patient Posttraumatic Stress Outcomes | 8-15 sessions of therapy or after 5 months since initial assessment, whichever comes first
  Patient posttraumatic stress symptom severity will be assessed via using the PTSD Symptom Scale - Interview, administered following referral to the study and after 8-15 sessions of therapy, or after 5 months since initial assessment, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Edna B Foa, Ph.D., Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Evans Army Community Hospital (EACH), Ft. Carson, Colorado Springs, Colorado
  - Blanchfield Army Community Hospital (BACH), Ft. Campbell, Fort Campbell North, Kentucky
  - William Beaumont Army Medical Center (WBAMC), Ft. Bliss, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foa EB, McLean CP, Brown LA, Zang Y, Rosenfield D, Zandberg LJ, Ealey W, Hanson BS, Hunter LR, Lillard IJ, Patterson TJ, Rosado J, Scott V, Weber C, Wise JE, Zamora CD, Mintz J, Young-McCaughan S, Peterson AL; STRONG STAR Consortium. The effects of a prolonged exposure workshop with and without consultation on provider and patient outcomes: a randomized implementation trial. Implement Sci. 2020 Jul 29;15(1):59. doi: 10.1186/s13012-020-01014-x. PMID 32727509